CLINICAL TRIAL: NCT02781636
Title: A European Trial to Assess the Efficacy of an Implantable Wireless Neuromodulation Device at the Tibial Nerve to Treat Urinary Urgency Incontinence
Brief Title: Protect Chronic Tibial Nerve Stimulator (CTNS) System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Replaced by US RCT
Sponsor: Uro Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30-00136
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Urge Incontinence
Keywords: Efficacy; Implantable; Wireless; Neuromodulation; Device; Tibial
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic Tibial Implant Arm (Experimental): StimGuard Protect System (Chronic Tibial Nerve Stimulation) Implant Procedure. Lead implanted adjacent to tibial nerve. Wireless rechargeable system.
  Interventions: Device: Device: StimGuard Protect System

INTERVENTIONS:
Device: Device: StimGuard Protect System — Lead implanted adjacent to tibial nerve. Wireless rechargeable system.
  Other Names: Chronic Afferent Nerve Stimulation

SUMMARY:
30 patient Study. All patients implanted with StimGuard Protect System. Patient followed out to 90 days.

DETAILED DESCRIPTION:
The proposed therapy is called chronic tibial nerve stimulation (CTNS), which is a low-risk, minimally invasive chronic implant for the treatment of urgency urinary incontinence. CTNS works by the same mechanism as percutaneous tibial nerve stimulation (PTNS), but is provided for chronic use with an implantable device. CTNS treatment involves the placement of a minimally invasive stimulator with an embedded receiver at the tibial nerve. The Protect CTNS System has an external transmitter that activates the implanted stimulator and sends mild electrical pulses to the tibial nerve. These impulses travel to the sacral nerve plexus, the group of nerves at the base of the spine responsible for bladder function. Since stimulation with the Protect CTNS System is chronic it is expected that bladder activity can be changed more quickly and without the frequency of treatments related to PTNS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder with urgency urinary incontinence

Exclusion Criteria:

* Primary complaint of stress urinary incontinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Urge Incontinence Episodes | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- UZA, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Upon Study Completion